CLINICAL TRIAL: NCT05722093
Title: Manzhi Guben Granules Improve Novel Coronavirus Infection (COVID-19) Efficacy and Safety of Convalescent Exercise Tolerance -- A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: MG Granules Improve COVID-19 Efficacy and Safety of Convalescent Exercise Tolerance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other); Suzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0094
Record Dates: First submitted 2023-02-08; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manzi Guben granules (Experimental): Administration cycle of Manzhi Guben granules: 1-4 weeks; Usage: 10g once, twice a day, washed with boiling water.
  Interventions: Drug: Manzi Guben granules
- placebo group (Placebo Comparator): Administration cycle of Manzhi Guben granules simulator: 1-4 weeks; Usage: 10g once, twice a day, washed with boiling water.
  Interventions: Drug: Manzi Guben granules

INTERVENTIONS:
Drug: Manzi Guben granules — Administration cycle of Manzhi Guben granules: 1-4 weeks; Usage: 10g once, twice a day, washed with boiling water.
  Other Names: test group

SUMMARY:
The global coronavirus pandemic has infected nearly 659 million people and killed more than 6.6 million in the past three years. The symptoms of in-hospital recovery are long and difficult after epidemiological infection of 2019-NCo5. 76% of the 1,733 discharged patients in Wuhan in 2020 still had at least one symptom of discomfort 6 months after infection, with fatigue or muscle weakness being the most common (63%). Foreign Research: In the United States, 15 percent of 16,091 people infected with COVID-19 in 2021 had symptoms that persisted two months after infection. Novel Coronavirus Infection Diagnosis and Treatment Protocol (Trial 10th Edition) For patients recovering from novel coronavirus infection, TCM syndrome differentiation can be carried out according to the Guidelines for Home-based TCM Intervention for Patients Infected with Novel Coronavirus, and appropriate TCM prescriptions should be given for intervention.

DETAILED DESCRIPTION:
In the past three years, the novel coronavirus pandemic has infected nearly 659 million people and caused more than 6.6 million deaths. Due to the continuous existence of the mutation of the novel coronavirus strain, the increased infectivity of the virus and the persistent immune escape potential of the virus, the number of patients infected with the novel coronavirus increased, and the infection peak followed. According to the latest information from the press conference of the Joint Prevention and Control Mechanism of The State Council, from December 8, 2022 to January 12, 2023, a total of 59,938 deaths related to novel coronavirus infection occurred in medical institutions across the country .

TCM has a history of thousands of years in the prevention and treatment of diseases and has accumulated rich clinical experience. For example, it is recorded in the Huangdi Neijing · Suwen that "the five epidemics are easy to be infected with each other, with no problem of size and similar symptoms". Written in the late Eastern Han Dynasty, Treatise on Febrile and Miscellaneous Diseases is a clinical masterpiece on the treatment of external febrile diseases, including most acute infectious diseases, and is known as the "ancestor of the book". By the Ming and Qing Dynasties, TCM had a more profound understanding of infectious diseases, formed a relatively complete theoretical system of febrile diseases, and made great achievements in the treatment of epidemics. In traditional Chinese medicine, the novel coronavirus infection epidemic is called "plague", "plague", "blight", etc., characterized by rapid onset and strong infectivity, middle-aged and elderly patients are often seriously ill, and some clinical symptoms are protracted and difficult to cure, which seriously affects the quality of life of patients . Domestic researchers conducted a follow-up study on 1,733 patients discharged from Wuhan Yintan Hospital between January 7 and May 29, 2020, and found that 76% of patients with novel coronavirus pneumonia still had at least one persistent symptom 6 months after the onset of the disease, with fatigue or muscle weakness being the most common (63%) [4]. Foreign researchers conducted a follow-up study on 16,091 adult patients with novel coronavirus in the United States from February 5, 2021 to July 6, 2022, and 15% of the patients reported persisting symptoms 2 months after infection [5]. Therefore, how to effectively delay symptoms and promote recovery is one of the key concerns in the research field of novel coronavirus infection.

Currently recognized effective drugs for the treatment of novel coronavirus, such as Paxlovid , Molnupiravir , Remdesivir , glucocorticoid, monoclonal antibody, etc., are mainly used to prevent high-risk patients with novel coronavirus infection from becoming severe or to reduce the fatality rate. However, there is still a lack of effective modern medical treatment for promoting body recovery and improving exercise tolerance.

New York Heart Association (NYHA) cardiac function scale, dyspnea scale and other measures to assess patients' activity ability, but such assessment measures are more dependent on patients' subjective feelings; Objective data evaluation has more clinical guiding value. The 6-minute walk test (6MWT) is simple, economical and safe, and can better reflect the exercise tolerance and cardiopulmonary function of patients. It is widely used to evaluate the efficacy and rehabilitation effect of patients with cardiovascular diseases and chronic respiratory diseases.

Although drugs can be used for symptomatic treatment such as cough and phlegm, there is no effective western medicine to relieve these symptoms such as fatigue, muscle weakness, qi promotion of sweat, fear of wind and cold, loss of appetite and other symptoms. Citing an article on the diagnosis and treatment of novel coronavirus published by Nature, a top international scientific journal, it is believed that at the current stage, active research and development of drugs that can alleviate symptoms of novel coronavirus infection, promote the recovery of the disease and improve the quality of life, as well as the diagnosis and treatment of mild to moderate novel coronavirus patients will have huge public health benefits [7]. Jade screen, as a famous prescription for the treatment of surface deficiency syndrome, comes from Wei Yilin's "Prescription for the effect of the World Medicine" in the Yuan Dynasty (some researchers also believe that it comes from Zhu Zhenheng's "Danxi Xin Method" in the Yuan Dynasty). The party has the beneficial effect of gas-solid table stop sweat, attending table is not solid, spontaneous perspiration evil wind, complexion white, pale tongue moss thin white, pulse vain, run-down cou justified is susceptible to the wind. The jade screen is made of Astragalus, fried white art and windproof. Astragalus is mainly used for spleen and lung Qi deficiency, which is used to benefit Qi and solid surface, and is the king medicine. White art invigorating spleen and qi, helping astragalus qi and solid surface, as minister medicine; Windproof table and wind evil, as a tonic.

However, there are few prospective clinical intervention studies on the use of Manzhi Guben granules for symptomatic supportive treatment during outpatient treatment of convalescent patients with novel coronavirus infection, and there is still a lack of high-quality clinical evidence-based medical evidence on its effectiveness in improving exercise tolerance of convalescent patients after novel coronavirus infection. This provides a good opportunity for the research of this project. By means of modern medical research, it is found that the main components of Manzhi Guben granules (Yupingfeng + Angelica sinensis) are: (1) Astragalus supplementing Qi and consolidating surface, antiviral infection, significant stimulation of interferon system, regulating and promoting humoral and cellular immunity; (2) Atractylodes atractylodes can nourish qi, invigorate spleen, dry dampness, enhance cellular and humoral immunity, and promote phagocytosis of macrophages; (3) Wind-proof and wind-dispelling, which can enhance immune function and fight infection; (4) Angelica sinensis: It has anti-thrombotic effect, improves blood circulation, improves coronary circulation in cardiovascular system, has anti-inflammatory and analgesic effect, lowers blood sugar effect, and has protective effect on lung. Some recent studies have found through modern pharmacological research means that a variety of active compounds in the prescription of Yupingfeng can play a role in the prevention and treatment of novel coronavirus infection through multi-target and multi-pathway [9,10], which further provides the basic theoretical basis for the clinical application of Manzhi Guben granules.

The research results of molecular mechanism of TCM prevention and treatment of novel coronavirus infection and clinical efficacy observation provide certain reference for the follow-up high-quality clinical research . The Research team has published an article in Pharmacological Research on the diagnosis and treatment of novel coronavirus infection : Analyzed in 2020 registered in the Chinese clinical trial registry of 130 intervention new coronavirus infection in clinical research of traditional Chinese medicine, found that: Single-center studies accounted for 60.8%, non-placebo controls for 86.2%, open-label or unstated blinds for 30.8% and 60.8%, and 80.8% of clinical studies enrolled no more than 300 patients. Therefore, high quality RCTs studies on the intervention of traditional Chinese medicine in patients with novel coronavirus infection can not only reflect the characteristics and advantages of traditional Chinese medicine, but also provide reliable clinical research results, which has become the main target of current research on the treatment of novel coronavirus infection by traditional Chinese medicine.

In summary, this study will closely focus on the effect of Manzhi Guben granules on improving exercise tolerance of patients with novel coronavirus during recovery period. A multicenter, randomized, double-blind, placebo-controlled high-quality clinical study was conducted to determine the efficacy and safety of Manzhi Guben granules in exercise tolerance recovery and symptom relief in patients infected with novel coronavirus. Finally, it will provide some reference for clinical and basic research on the treatment of novel coronavirus infection by Chinese patent medicine and the promotion of patients' recovery. Ii. Overall Objectives of the Project

To evaluate the effectiveness and safety of Manzhi Guben granules in improving exercise tolerance and promoting body rehabilitation in patients with novel coronavirus infection. To provide reliable evidence support for the treatment and improvement of novel coronavirus infection with Manzhi Guben granules.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic criteria for convalestion-phase of COVID-19 patients: Patients with COVID-19 have entered the convalestion-phase when they meet any of the following criteria and other symptoms improve: 1) two consecutive negative nucleic acid tests with Ct values ≥35; 2) The antigen test results were negative for three consecutive days; 3) After staying at home for 7 days, the fever has subsided for more than 24 hours without using antipyretic drugs; (2) Middle-aged and elderly outpatients aged 50-80 (including 50 and 80 years old), regardless of gender; (3) The main clinical manifestations were fatigue, shortness of breath, cough (satisfying at least two main symptoms), and the results of 6-minute walking test were less than 80% of the predicted value (about 450-500 meters); Can be accompanied by poor puppie full, loose stool, light fat tongue, thin white or thin greasy moss, pulse floating, the performance of lung qi deficiency. (4) Voluntarily participate in this clinical study, give informed consent and sign informed consent.

Exclusion Criteria:

1. Severe and critically ill hospitalized patients with novel coronavirus infection; (2) accompanied by tumor, immune deficiency disease; (3) The researcher thinks that it is not appropriate to participate in this clinical research; (4) Suspected or confirmed history of alcohol and drug abuse; (5) Known or suspected allergic history to the study drug and its excipients; (6) participated in other clinical investigators within 3 months before screening; (7) Patients with severe neurological, cardiac, pulmonary, hematopoietic, endocrine, musculoskeletal motor system and other primary diseases and mental disorders; (8) Patients with clinical manifestations of Yin deficiency and fire flourishing (red tongue and thin pulse) or phlegm-dampness and lung stagnation (white and greasy moss, slippery pulse strings); (9) Life expectancy is less than 12 weeks due to underlying diseases.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Results of 6 min walking test on day 14 | 14 days
  Results of 6 min walking test on day 14 after treatment

SECONDARY OUTCOMES:
Results of 6 min walking test on the 28 | 28 days
  Results of 6 min walking test on the 28th day after treatment
Pulmonary ventilation function on day 14 and 28 | 14 days and 28 days
  Pulmonary ventilation function on day 14 and 28 after treatment

CONTACTS AND LOCATIONS:
Overall Officials: yongan xu, doctor, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University